CLINICAL TRIAL: NCT04364386
Title: Feasibility Clinical Investigation Using the InPress Device for the Treatment of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alydia Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P-001
Record Dates: First submitted 2020-02-20; First posted 2020-04-28 (Actual); Results first posted 2023-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Post Partum Hemorrhage
Keywords: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- InPress (Experimental): Treatment with InPress Device for Postpartum Hemorrhage
  Interventions: Device: InPress Device

INTERVENTIONS:
Device: InPress Device — Treatment with InPress Device for Postpartum Hemorrhage

SUMMARY:
Feasibility trial of the InPress Device to treat postpartum hemorrhage (PPH).

DETAILED DESCRIPTION:
10 subjects in first in woman trial with ethics committee oversight. Women who developed postpartum hemorrhage were treated with the InPress Device. The intent of treatment was to quickly reduce or stop blood flow by addressing the driving cause of hemorrhage: uterine atony.

The primary objective is to verify the safety of the InPress Device in humans, including: 1. Absence of SAEs related to the use of the InPress Device intra- and post-procedure. 2. Evaluate any observable damage of the uterus, cervix, or vagina due to the use of the InPress Device. 3. Evaluate occurrence of uterine inversion or folding during the use of the InPress Device.

The secondary objectives include evaluations of: 1. Ability to easily place the InPress Device transvaginally. 2. Ability to connect the InPress Device to vacuum and maintain desired negative pressure. 3. Ability of InPress Device to contract the uterus to a level that reduces or stops blood loss and avoids further surgical intervention. 4. Evaluate time from insertion and start negative pressure to visible reduction of blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Subject or her legally authorized representative is able to understand and provide consent to participate in the clinical investigation
* Female adult subjects (>18 years of age)
* Subjects who present with an atonic uterus for at least 10 minutes after expulsion of placement with failure to obtain contraction and/or Subjects who have lost blood post-partum >= 500 ml and according to the Investigator's judgment, require an intervention.

Exclusion Criteria:

* Subjects who do not provide informed consent to participate in the clinical investigation.
* Subjects who deliver at a uterus size < 34 weeks.
* Subjects who have lost greater than 1000 ml of blood.
* Subjects who have abnormal PT, PTT and INR
* Subjects who present with retained placenta, uterine lacerations, or for any other conditions outside of atonic post-partum hemorrhage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who have just delivered a baby.
Enrollment: 10 (Actual)
Dates: Start 2014-07-27 (Actual); Primary Completion 2015-02-11 (Actual); Study Completion 2015-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuditiya Purwosunu, MD, Principal Investigator — Indonesia University
Locations (2):
- Indonesia (2):
  - Dr. Cipto Mangunkusumo Hospital, Jakarta
  - RSIA Budi Kemuliaan Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No
No plan.

REFERENCES:
- [Result] Purwosunu Y, Sarkoen W, Arulkumaran S, Segnitz J. Control of Postpartum Hemorrhage Using Vacuum-Induced Uterine Tamponade. Obstet Gynecol. 2016 Jul;128(1):33-36. doi: 10.1097/AOG.0000000000001473. PMID 27275795

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | InPress
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | InPress
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Indonesia | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Related SAE
Description: Number of device related SAEs
Time Frame: 6 weeks
Measure: Number; unit: SAEs
Arm/Group | InPress
Number analyzed (Participants) | 10
SAEs | 0

2. Primary Outcome: Number of Participants With Damage to Cervix, Uterus or Vagina
Description: Number of any observable damage to cervix, uterus, vagina
Time Frame: During the procedure
Measure: Number; unit: participants
Arm/Group | InPress
Number analyzed (Participants) | 10
participants | 0

3. Primary Outcome: Number of Participants With Uterine Inversion or Folding
Description: Number of uterine inversion or folding during procedure
Time Frame: During the procedure
Measure: Number; unit: participants
Arm/Group | InPress
Number analyzed (Participants) | 10
participants | 0

4. Secondary Outcome: Number of Participants With User Feedback on Placement of InPress
Description: Positive user feedback on placement transvaginally
Time Frame: During the procedure
Measure: Number; unit: participants
Arm/Group | InPress
Number analyzed (Participants) | 10
participants | 10

5. Secondary Outcome: Number of Participants With User Feedback on Connection to Vacuum
Description: Positive user feedback on connection to vacuum and maintenance of desired negative pressure
Time Frame: During the procedure
Measure: Number; unit: participants
Arm/Group | InPress
Number analyzed (Participants) | 10
participants | 9

6. Secondary Outcome: Time to Uterine Contraction
Description: Time to uterine contraction to a level that reduces or stops blood flow. Duration is exactly between 1 and 2 minutes for 1 participant, while the available data only suggests that it was less than 2 minutes for the rest of the participants but the exact duration cannot be narrowed down to 1-2 minutes.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | InPress
Number analyzed (Participants) | 10
Participants
  1-2 minutes | 1
  Less than 2 minutes | 9

7. Secondary Outcome: Time
Description: Time from insertion to removal of the device
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | InPress
Number analyzed (Participants) | 10
minutes | 152 (111.7)

ADVERSE EVENTS:
Arm/Group | InPress
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InPress (N=10)
urine retention post extraction with forceps with infected opened perineal laceration (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No